CLINICAL TRIAL: NCT04523922
Title: Oxytocin to Enhance Integrated Exposure-Based Treatment of Co-occurring Alcohol Use Disorder and PTSD
Brief Title: Oxytocin to Enhance Integrated Treatment for AUD and PTSD
Acronym: COPE+OT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sudie Back, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00103198
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: PTSD; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin Treatment Group (Experimental): Participants will receive 12 weekly sessions of Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure (COPE Therapy), plus intranasal Oxytocin.
  40-IU dose of Oxytocin self-administered 30 minutes prior to the start of each weekly COPE session.
  Interventions: Drug: 40 IU Intranasal Oxytocin; Behavioral: Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure
- Placebo Group (Active Comparator): Participants will receive 12 weekly sessions of Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure (COPE Therapy), plus placebo (intranasal saline spray).
  Intranasal dose of saline spray self-administered 30 minutes prior to the start of each weekly COPE session.
  Interventions: Drug: Placebo; Behavioral: Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure

INTERVENTIONS:
Drug: 40 IU Intranasal Oxytocin — 40 IU Intranasal Oxytocin self administered 30 minutes prior to each COPE session.
  Other Names: oxytocin
  Arms: Oxytocin Treatment Group
Drug: Placebo — Placebo (intranasal saline spray) self administered 30 minutes prior to each COPE session.
  Other Names: saline
  Arms: Placebo Group
Behavioral: Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure — 12 weekly sessions of COPE therapy for PTSD and AUD.
  Other Names: COPE

SUMMARY:
The primary objective of the proposed Stage II study is to examine the efficacy of oxytocin (OT) as compared to placebo in reducing (1) alcohol use disorder (AUD) symptoms, and (2) post-traumatic stress disorder (PTSD) symptoms among Veterans receiving COPE therapy (Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure). To evaluate purported neurobiological mechanisms of change, we will employ functional magnetic resonance imaging (fMRI) at pre- and post-treatment.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD) frequently co-occur and are associated with significant morbidity, mortality, and health care expenditures. Military Veterans are at increased risk for co-occurring AUD and PTSD, with prevalence rates 2-4 times higher than the general population. Our group developed an integrated intervention entitled Concurrent Treatment of PTSD and Substance Use Disorders using Prolonged Exposure (COPE). COPE incorporates empirically validated cognitive-behavioral techniques for AUD with Prolonged Exposure (PE) therapy for PTSD. Several randomized controlled trials among Veterans and civilians demonstrate efficacy of COPE in significantly reducing AUD and PTSD symptoms. Despite the positive findings, there remains substantial room for improving treatment outcomes and enhancing retention. Accumulating data suggest that the neuropeptide oxytocin (OT) is a promising candidate to enhance psychosocial interventions for co-occurring AUD and PTSD, as OT targets neurobiological and behavioral dysregulation common to both disorders. Preclinical and clinical studies demonstrate the ability of OT to ameliorate a variety of alcohol-related behaviors (e.g., craving, withdrawal symptoms, tolerance, ethanol self-administration), enhance fear extinction, and promote prosocial behaviors associated with successful psychosocial treatment outcomes. In a randomized controlled pilot study, our group found that OT administration prior to weekly Prolonged Exposure (PE) therapy sessions was safe, well-tolerated, and resulted in accelerated reduction in PTSD symptoms as compared to placebo. Although the empirical and theoretical support for augmenting psychosocial interventions such as COPE with OT is robust, no studies to date have examined this combined approach. The primary objective of the proposed Stage II study is to examine the efficacy of OT as compared to placebo in reducing (1) AUD symptoms, and (2) PTSD symptoms among Veterans (50% women) receiving COPE therapy. To accomplish this, we will employ a manualized, evidence-based, cognitive-behavioral intervention (COPE); a randomized, double-blind, placebo-controlled study design; and standardized, repeated dependent measures of clinical outcomes at multiple time points. In addition, to investigate neurobiological mechanisms of change, we will employ functional magnetic resonance imaging (fMRI) at pre-and post-treatment .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; U.S. military Veteran, any race or ethnicity; aged 18-70 years.
2. Able to provide written informed consent.
3. Meet DSM-5 diagnostic criteria for current moderate to severe alcohol use disorder.
4. Meet DSM-5 diagnostic criteria for current PTSD as assessed by the CAPS-5.
5. Participants may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria) or anxiety disorders. Concurrent substance use disorders (e.g., marijuana) are acceptable provided alcohol is the participant's primary substance of choice.
6. Participants taking psychotropic medications will be required to be maintained on a stable dose for at least 4 weeks before study initiation.

Exclusion Criteria:

1. Meeting DSM-5 criteria for a history of or current psychotic or bipolar affective disorders, or with current suicidal or homicidal ideation and intent. Those participants will be referred clinically for services.
2. Participants on psychotropic medications which have been initiated during the past 4 weeks.
3. Acute alcohol withdrawal as indicated by CIWA-Ar scores >8.
4. Pregnancy or breastfeeding for women.
5. For MRI scan component: history of seizures or severe head injury, implanted metal devices or other metal (e.g., shrapnel). These participants will be eligible to enroll in the clinical trial but will not be eligible to participate in the neuroimaging component of the study.
6. Currently enrolled in behavioral treatment for AUD or PTSD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol use | From baseline to week 12 and 3 and 6 month follow ups
  Change in percent days abstinent and heavy drinking days as measured by the TimeLine Follow-Back (TLFB).
Change in PTSD symptom severity - clinician rated | From baseline to week 12 and 3 and 6 month follow ups
  Change in clinician-rated PTSD symptom severity will be measured with the Clinician Administered PTSD Scale for DSM-5 (CAPS-5).
Change in PTSD symptom severity - self report | From baseline to week 12 and 3 and 6 month follow ups
  Change in self-reported PTSD symptom severity will be measured with the PTSD Checklist for DSM-5 (PCL-5).

CONTACTS AND LOCATIONS:
Overall Officials: Sudie Back, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Back SE, Flanagan JC, Killeen T, Saraiya TC, Brown DG, Jarnecke AM, Rothbaum AO, Joseph J, Ana ES, de Arellano A, Shoemaker HL, Dixon RA, Nietert PJ, Brady KT. COPE and oxytocin for the treatment of co-occurring PTSD and alcohol use disorder: Design and methodology of a randomized controlled trial in U.S. military veterans. Contemp Clin Trials. 2023 Mar;126:107084. doi: 10.1016/j.cct.2023.107084. Epub 2023 Jan 13. PMID 36646315